CLINICAL TRIAL: NCT04603222
Title: Evaluation of SUMMIT BRUSH in Treatment of Blepharitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Giles Duffield, Principal Investigator, University of Notre Dame
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUMMIT BRUSH
Record Dates: First submitted 2020-10-19; First posted 2020-10-26 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-10

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Intervention Model Description: This multi-site study will involve 60 subjects. Each site will have 20 participants. Each site will divide participants into two groups of 10. The control group will receive the standard of care. The standard of care would be Ocusoft Lid Scrub Original Foaming Eyelid Cleanser to be used once per day. The treatment group would receive the same treatment as the control group with the addition of the experimental disposable ocular brush. The foam will be applied to the brush and the subjects will gently provide a scrubbing action to the eyelids while keeping the eyelids closed. They will also be instructed to perform treatment once per day and to dispose of the brush after two weeks and replace it with a new brush.
  Each participant will be asked to return to their respective site for two follow up visits. The first visit will take place at two weeks commencing treatment and the final visit will take place two weeks later for a total treatment duration of one month.
Who Masked: Outcomes Assessor
Masking Description: All SPEED scores and digital images would then be de-identified to avoid any bias by the principal investigator and his research staff.
  These scores and images would be uploaded and sent electronically via encrypted password protected file to Giles Duffield, PhD. for interpretation and statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Group treating blepharitis with SUMMIT BRUSH and Ocusoft Lid Scrub Original Foaming Eyelid Cleanser once a day
  Interventions: Device: SUMMIT BRUSH; Other: Ocusoft Lid Scrub Original Foaming Eyelid Cleanser
- Control Group (Active Comparator): Group treating blepharitis with Ocusoft Lid Scrub Original Foaming Eyelid Cleanser once a day
  Interventions: Other: Ocusoft Lid Scrub Original Foaming Eyelid Cleanser

INTERVENTIONS:
Device: SUMMIT BRUSH — SUMMIT BRUSH used for the treatment of blepharitis
  Arms: Treatment Group
Other: Ocusoft Lid Scrub Original Foaming Eyelid Cleanser — treating blepharitis with Ocusoft Lid Scrub Original Foaming Eyelid Cleanser

SUMMARY:
Dry Eye Disease (DED) is a multifactorial disease that affects ~15-30 million people in the USA alone. It creates an enormous societal and economic burden, decreases productivity in the workplace, and affects the quality of lives of the people affected by this disease. DED is primarily caused by blepharitis, a chronic inflammation of the eyelid margins. If left untreated, blepharitis results in the obstruction and loss of the glands responsible for tear film production. The standard of care is the use of self-administered at home commercially available products, e.g., eyelid foams, gels, and pads. Although these products are helpful, they have limitations. Patients often require expensive in office procedures, e.g., lid debridement with exfoliation devices or more expensive procedures. The scope of this project is to evaluate the effectiveness of a new self-administered disposable ocular brush used in conjunction with the most common eyelid cleanser. The investigators are looking to see if combining the microexfoliation provided by the brush with the eyelid cleanser is more effective at removing the eyelid debris than the cleanser alone.

DETAILED DESCRIPTION:
Dry Eye Disease is a multifactorial disease that affects approximately 15-30 million people in the United States alone. it creates an enormous societal and economic burden, decreases productivity in our workplace, and significantly affects the quality of lives of the people affected by this disease. Appoximately 86% of Dry Eye Disease is caused by Blepharitis, a chronic inflammation of the eyelid margins. If left untreated, Blepharitis results in the obstruction and eventual loss of the glands responsible for a critical component of tear film production.

The standard of care in the treatment of Blepharitis is the use of self administered at home commercially available products such as eyelid foams, gels, and pre moistened pads. These products contain non abrasive cleansers designed to remove the buildup of biofilm and excess microorganisms on the lid margin. Although these products are helpful, they do have some limitations. Many patients still require more expensive in office procedures such as lid debridement with electro-mechanical exfoliation devices or other even more expensive procedures.

The scope of this project is to evaluate the effectiveness of a new self administered disposable ocular brush used in conjunction with the most commonly prescribed commercially available eyelid cleanser. The investigators are looking to see if combining the microexfoliation provided by the brush with the eyelid cleanser is more effective at removing the eyelid debris (scurfs, collarettes, and demodex) than the cleanser alone.

Hypothesis: The Summit Ocular Brush used in conjunction with Ocusoft Original lid cleanser is more effective than the cleanser alone at removing the debris (scurfs, collarettes, and demodex) from the eyelids in the treatment and management of Blepharitis.

The investigators want to determine if the addition of the ocular brush with the eyelid cleanser has synergistic effects on reducing the signs and symptoms of Blepharitis and Dry Eye Disease. They also hope to learn that with this additional step, further and more expensive procedures could be avoided thereby decreasing the overall economic burden on the patient and society as a whole.

Recruitment of participants: Dr. Kevin Danahey, Dr. Richard Mangan, and Dr. Paul Karpecki are the three clinical investigators for this multi-site study. They are all directors of Dry Eye Clinics and regularly see patients throughout the course of the day. Potential participants will be identified during routine office visits. Participants will be identified by subjective symptoms and objective signs of Blepharitis. The SPEED (Standardized Patient Evaluation of Eye Dryness) Questionnaire will be utilized to identify symptoms and Slit Lamp Biomicroscopy will be used to identify objective clinical signs of Blepharitis. Once patients are identified as potential candidates, they will be informed by the investigator that they are a candidate for a study and asked if they would be interested in participating. A brief explanation of the study will be given and the patient will be informed that regardless of which group they are assigned to, they would still be receiving the current standard of care. The candidates would then be asked to return so that the Investigators may provide informed consent, thorough written and verbal instructions, HIPPA forms, SPEED questionnaires, and treatment products. The patients would also have digital photos and video performed with Slit Lamp Biomicroscopy at that time. These images would only involve the lids and lashes of the subjects allowing the investigators to protect the identity, gender, and age of the subject.

Study: This multi-site study will involve 60 subjects. Each site will have 20 participants. Each site will divide participants into two groups of 10. The control group will receive the standard of care. The standard of care would be Ocusoft Lid Scrub Original Foaming Eyelid Cleanser to be used once per day. The treatment group would receive the same treatment as the control group with the addition of the experimental disposable ocular brush. The foam will be applied to the brush and the subjects will gently provide a scrubbing action to the eyelids while keeping the eyelids closed. They will also be instructed to perform treatment once per day and to dispose of the brush after two weeks and replace it with a new brush.

Each participant will be asked to return to their respective site for two follow up visits. The first visit will take place at two weeks commencing treatment and the final visit will take place two weeks later for a total treatment duration of one month. During each visit, the subjects will fill out the SPEED questionnaire and digital images and videos will be taken. The length of each visit should take no longer than 15 minutes. At the conclusion of the study, subjects in the treatment group will be asked to discontinue the experimental brush. They would be asked to continue with the current standard of care.

All SPEED scores and digital images would then be de-identified to avoid any bias by the principal investigator and his research staff. These scores and images would be uploaded and sent electronically via encrypted password protected file to Giles Duffield, PhD. for interpretation and statistical analysis.

Anterior blepharitis is an ophthalmologic condition characterized by an inflammation of the eyelid margins. It can be acute or chronic with chronic being the more common form. Blepharitis is a clinical diagnosis based on irritation of the lid margins with flaking and crusting of the lashes.

The main treatment for blepharitis is good eyelid hygiene and elimination of triggers that exacerbate symptoms (Pflugfelder SC, Karpecki PM, Perez VL. Treatment of blepharitis: recent clinical trials. Ocul Surf. 2014 Oct;12(4):273-84).

Blepharitis is not specific to any group of people. It affects people of all ages, ethnicities, and gender. It is more common in individuals older than the age of 50. The total number of cases in the US at any one time is not known. In a 2009 US survey, 37% of patients seen by an ophthalmologist and 47% of patients seen by an optometrist had signs of blepharitis.

The exact pathophysiology of blepharitis is not known. The cause is most likely multifactorial. Causative factors include a combination of chronic low-grade bacterial infections of the ocular surface, inflammatory skin conditions such as atopy and seborrhea, and parasitic infestations with Demodex mites.

There are a number of products on the market that aid in reducing the inflammatory and bacterial load to the lid margin and lashes. However, mechanical debridement (or lid scrubs) is best at removing debris and the bacterial biofilm that forms in chronic cases. As one ages, near vision and dexterity worsens. Timely and appropriate lid hygiene then suffers that may result in lid and ocular infection, as well as vision loss.

The Summit Ocular Brush proposed here should improve the effectiveness of personal home lid hygiene, even in an aging population. This is what the Investigators wish to study.

The experimental design includes one experimental group and one control group. Subjects will be divided up such that each clinic collects 10 subjects from each group. This will provide us with 30 experimental and 30 control subjects and spread evenly between the three separate clinical locations. Data analysis will be of still images taken from video and photographic images of the eye lid margins.

Data will be in the form of counts of eyelid debris, specifically 1) scurfs, 2) collarettes, and 3) demodex. Analysis will be performed by Dr. Duffield and his team at the University of Notre Dame and will be performed blind. Each subject data set will only be identifiable by a code, which will not allow for prior knowledge of origins of treatment group. The n=30 sample size is deemed appropriate for the application of standard statistical methods on continuous data, specifically parametric t-test or non-parametric Mann-Whitney test. Analysis at the subgroup level (with 3+ groups), such as incorporation of gender or age fractionation, parametric ANOVA or nonparametric Kruskal-Wallis tests will be performed on the data, followed by post-hoc pair wise comparison tests. In all cases, alpha will be set at 0.05, i.e. p< 0.05 will be seemed significant. The relatively large sample size of 30 subjects in each main group affords us the opportunity to examine subgroup affects without concern that the Investigators have insufficient numbers of subjects.

Lid Scrubs are listed at every stage of the treatment algorithm for anterior blepharitis. As patients age, their ability to perform proper lid scrubs / hygiene declines. Without proper mechanical debridement of lid and lash flakes, scurfs, collarettes, or mites, this condition can remain chronic or recalcitrant. Chronic use of topical antibiotics promotes bacterial resistance and chronic use of steroids puts patients at risk for infection and elevated intra-ocular pressure. With sound and proper debridement technique using the Summit Ocular Brush, this should lesson the need for such prescription medication.

Patients will be followed by their doctor's normal standard of care protocol.

The experimental design includes one experimental group and one control group.

Subjects will be divided up such that each clinic collects 10 subjects from each group. This will provide us with 30 experimental and 30 control subjects and spread evenly between the three separate clinical locations. Data analysis will be of still images taken from video and photographic images of the eye lid margins. Data will be in the form of counts of eyelid debris, specifically 1) scurfs, 2) collarettes, and 3) demodex. Analysis will be performed by Dr. Duffield and his team at the University of Notre Dame and will be performed blind. Each subject data set will only be identifiable by a code, which will not allow for prior knowledge of origins of treatment group. The n=30 sample size is deemed appropriate for the application of standard statistical methods on continuous data, specifically parametric t-test or non-parametric Mann-Whitney test. Analysis at the subgroup level (with 3+ groups), such as incorporation of gender or age fractionation, parametric ANOVA or nonparametric Kruskal-Wallis tests will be performed on the data, followed by post-hoc pair wise comparison tests. In all cases, alpha will be set at 0.05, i.e. p< 0.05 will be seemed significant. The relatively large sample size of 30 subjects in each main group affords us the opportunity to examine subgroup affects without concern that the Investigators have insufficient numbers of subjects.

Patients will be followed by their doctor's normal standard of care protocol. Participants can be both male and female over the age of 18 with clinical signs and symptoms of Blepharitis (Staphylococcal and Demodex). Participants must exhibit visible collarettes, clear sleeves, and scurfs on the eyelid margins upon Slit Lamp Biomicroscopy.

Participants both male and female under the age of 18. Patients with any active hordeolum (stye), chalazion, periorbital cellulitis, or any evidence of allergic eyelid dermatitis. Participants will also be excluded if they have any active acute bacterial conjunctivitis or any active open periorbital wounds.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of blepharitis (Staphylococcal and Demodex).
* Must exhibit visible collarettes, clear sleeves, and scurfs on the eyelid margins upon Slit Lamp Biomicroscopy.

Exclusion Criteria:

* Hordeolum
* Chalazion
* Periorbital cellulitis
* Allergic eyelid dermatitis.
* Acute bacterial conjunctivitis
* Open periorbital wounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-10-24 (Estimated); Study Completion 2022-07-18 (Estimated)

PRIMARY OUTCOMES:
Change in blepharitis severity on eye lid margins | Initial visit, 2 week follow up, and 4 week follow up
  Digital photography will be used to asses the eye lid margins pre-treatment, during treatment, and post-treatment. The number of collarettes on the eyelashes will be counted at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Giles E Duffield, Ph.D., Principal Investigator — University of Notre Dame
Locations (3):
- United States (3):
  - University of Colorado, Boulder, Colorado
  - Michiana Eye Center, Mishawaka, Indiana
  - Kentucky Eye Institute, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No